CLINICAL TRIAL: NCT05617560
Title: Hospital@Home: Telemedical Care After Inpatient Hospital Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Innosuisse - Swiss Innovation Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-01440; am22Eckstein2
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Telemedicine
Keywords: Medgate; Patient transfer path; Telemedical care; Telephone consultation; Videocall consultation; ergebnisorientiertes Patientenassessment - AcuteCare (ePA-AC); Patient-Reported Experience Measures Survey (PREMS); Patient Reported Outcome Measures Survey (PROMS)

STUDY DESIGN:
Intervention Model Description: investigator-initiated, prospective, single-center clinical intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedical care (Experimental)
  Interventions: Other: Telemedical care

INTERVENTIONS:
Other: Telemedical care — Telemedical care will be provided to all participants after stationary hospital stay. This care will be in form of telephone consultations and / or videocall consultations with a medical physician. Depending on the individual medical history and the planned aftercare and procedure of the participants it will comprise of one or more such telephone consultations.

SUMMARY:
This pilot study is to investigate a patient transfer path from the hospital to Hospital@Home to their general practitioners (GPs) using telemedical procedures. Telemedical support will be executed by Medgate who will refer the patients to their GPs after the telemedical consultations are completed. Inclusion criteria is the need for short time follow up procedures that can be handled by telemedicine. Throughout the study, patient and stakeholder satisfaction will be measured and data-based methods will be developed to assess patient transfer success. Overall, new information flow and communication between the stakeholders (hospital, telemedicine and general practitioners) are defined and tested. The Hospital@Home pilot study is intended to become a flagship project for new healthcare models.

DETAILED DESCRIPTION:
This pilot study is to investigate a patient transfer path from the hospital to Hospital@Home to their general practitioners (GPs) using telemedical procedures.

The following study procedures are depicted:

Visit 1 (screening): Patients provide the name of their GP, the means of transport that they usually take to him, demographic data, past medical history and current medications.

The study team contacts the GP afterwards by phone to get his/her consent. The study team informs Medgate about the participant and the procedure. Next to that it will link Medgate technically to the case of the patient that Medgate can see the patient's documentation in the University Hospital Basel (USB) -ePortal.

Visit 2 (transfer): Before leaving the hospital, the participant will be instructed by a member of the study team on how and when to fill out the questionnaires. At this time, the participant and the USB physician will answer the first one. After Medgate has received the information from USB that the patient has been included in the study and has left the hospital, the patient will be contacted by Medgate and the appointment for the first teleconsultation will be made according to information from USB. The patient will be called by Medgate physician at the agreed time and the teleconsultation will be performed. Depending on the patient's condition and health status, further appointments are scheduled. The patient has the possibility to contact Medgate at any time (24/7) in case of an urgent medical matter. The patient receives the physician's recommendations in written form after each teleconsultation as their treatment plan via app or e-mail.

Visit 3...x (telecare): In advance of the first consultation via Medgate, the Medgate physician will log in into the USB-ePortal to get all important medical information about the patient. After that consultation the patient and the Medgate physician will answer a questionnaire. Depending on the clinical condition, health status and from this resulted procedure, the participant will be contacted several times. After the last consultation the Medgate physician will answer a questionnaire and will refer the patient back to the GP. The documentation will be sent to the GP and the USB. The GP will get a questionnaire as well.

Visit 4 (follow-up): On day x after the last consultation via Medgate the GP and the participant will answer the last questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent as documented by signature from the patient
* Planned hospital discharge
* Intended follow-up care, that is manageable with telemedicine

Exclusion Criteria:

* Significant mental or cognitive impairment
* Unable or not willing to sign informed consent
* Unable to understand German
* No possibility of telecommunication or use of such (app or phone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in PROMS (patient-reported outcome measures survey) | From Visit 2 (Transfer) up to Visit 4 (Follow up), approx. 2 weeks
  PROMS (patient-reported outcome measures survey): measure to asses a patient's quality of life affected by state of health. 6 standardized questions for self-assessment of the patient's state of health by the patient. The content of the questions relates to mobility, self-care, general activities, pain, anxiety and health in general. Questions are answered using Likert scales and qualitative free text answers. Scoring: 5 multiple choice questions (example pain: no pain, mild -, moderate -, severe -, extreme pain); (example general health: Scale from 0 - 100 (0 = worst health, 100 = best health imaginable)).
PREMS (patient reported experience measure survey) conducted by patients | From Visit 2 (Transfer) up to Visit 4 (Follow up), approx. 2 weeks
  PREMS (patient reported experience measure survey): satisfaction related questionnaire. Questions are answered using Likert scales (Format: 1: You completely disagree with this statement. 2: - not to. 3: - rather not to. 4: - neither accept nor reject them. 5: - a little too. 6: - majority to 7: You very much agree with this statement)
PREMS (patient reported experience measure survey) conducted by physicians | From Visit 2 (Transfer) up to Visit 4 (Follow up), approx. 2 weeks
  PREMS (patient reported experience measure survey): satisfaction related questionnaire. Questions are answered using Likert scales (Format: 1: You completely disagree with this statement. 2: - not to. 3: - rather not to. 4: - neither accept nor reject them. 5: - a little too. 6: - majority to 7: You very much agree with this statement)

OTHER OUTCOMES:
Change in self-care index (Selbstpflegeindex (SPI)) | From Visit 1 (Screening) up to Visit 3 (Telecare), approx. 1 week
  The SPI shows the need for care in each patient. The SPI ranges from values between 0 - 40, whereas a low SPI corresponds to more extensive need for care. It is the numeric score outcome of the ePA-AC, which is calculated from 10 ePA-AC questions.
Change in result-oriented patient assessment (ergebnisorientiertes Patientenassessment - AcuteCare (ePA-AC)) | From Visit 1 (Screening) up to Visit 2 (Transfer) assessed daily at the hospital, approx. 1 week
  The ePA-AC is focused on the nursing process and sub classifies activities of daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, Prof. Dr. med., Principal Investigator — University Hospital Basel, Division of Internal Medicine
Locations (1):
- University Hospital Basel, Division of Internal Medicine, Basel, Switzerland